CLINICAL TRIAL: NCT03490669
Title: A Phase 1 Multicenter, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Antitumor Activity of MSC-1 in Patients With Advanced Solid Tumors
Brief Title: Study to Evaluate Safety, PK, PD, Immunogenicity & Antitumor Activity of MSC-1 in Patients With Adv Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MSC-1-101; 2017-003320-79 (EudraCT Number)
Record Dates: First submitted 2018-02-07; First posted 2018-04-06 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors; Pancreatic Cancer; Non Small Cell Lung Cancer; Ovarian Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Multiple dose levels of MSC-1 treatment once every 3 weeks
  Interventions: Biological: MSC-1
- Dose Expansion (Experimental): MSC-1 treatment at the recommended Phase 2 dose once every 3 weeks
  Interventions: Biological: MSC-1

INTERVENTIONS:
Biological: MSC-1 — humanized monoclonal antibody for intravenous administration

SUMMARY:
This is a 2-part study to evaluate the safety and antitumor activity of MSC-1. MSC-1 is a first-in-class, humanized monoclonal antibody (IgG1) which binds to the immunosuppressive human cytokine Leukemia Inhibitory Factor (LIF), and is intended to treat adult patients with Advanced Solid Tumors.

In part 1, multiple dose levels of MSC-1 in patients with advanced solid tumors will be studied to determine the recommended dose for further evaluation of safety and efficacy in Part 2.

DETAILED DESCRIPTION:
MSC-1 is a first-in-class, humanized monoclonal antibody (IgG1) which binds to the immunosuppressive human cytokine Leukemia Inhibitory Factor (LIF), and is intended to treat adult patients with advanced solid tumors. LIF is a pleiotropic cytokine involved in many physiological and pathological processes including the promotion of an immunosuppressive environment. In cancer, it is hypothesized that LIF expressing malignancies co-opt this activity, creating an immunosuppressive tumor microenvironment as well as promoting the activity of cancer-initiating cell(s) (CICs). LIF is highly expressed in a subset of tumors across multiple solid tumor types.

During dose escalation, patients with advanced solid tumors will be treated with MSC-1 with the primary objective of determining the safety and tolerability of MSC-1 and defining an appropriate dose for further evaluation in dose expansion. MSC-1 will be administered intravenously (IV) until disease progression, unmanageable toxicity, withdrawal of consent or study termination.

In dose expansion, up to 4 parallel cohorts of patients with LIF-High tumors (NSCLC, Ovarian Cancer, Pancreatic Cancer), and a cohort of mixed solid tumors (referred to as the "basket cohort"), may be treated at the recommended expansion dose to further characterize the safety, tolerability, PK, PD and anti-tumor activity of MSC-1.

ELIGIBILITY:
Inclusion Criteria (All patients):

* Confirmed Advanced Unresectable Solid Tumor
* Measurable disease by RECIST 1.1 by CT or MRI
* Documented disease progression on or following last line of therapy
* Archival tumor sample for submission
* ECOG performance status 0 or 1
* Resolution of all acute, reversible toxic effects of prior therapy or surgical procedures to at least grade 1 (except alopecia and peripheral neuropathy to at least grade 2)
* Adequate organ function
* A limited number of patients enrolled in Dose Escalation may be required to agree to pre- and on-treatment tumor biopsies

Inclusion Criteria (Dose Expansion patients only)

* LIF- High NSCLC, Ovarian Cancer, or Pancreatic Cancer for the tumor-specific cohorts or Advanced Solid Tumor for the basket cohort as assessed by tumor tissue evaluation by IHC
* All patients enrolled in Dose Expansion must agree to undergo pre- and on-treatment tumor biopsies

Exclusion Criteria (All Patients):

* Systemic anti-cancer therapy within 4 weeks or 5 half-lives prior to study entry
* Previous or concurrent malignancy that could affect compliance with protocol or interpretation of results
* Clinically significant, unstable cardiovascular or pulmonary disease as specified in detail in the study protocol
* History of acquired or congenital immunodeficiency syndrome or receiving immunosuppressive therapy
* Uncontrolled infections or serologically positive HIV or hepatitis B or C infection
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or interfere with interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of MSC-1 and determine the recommended dose for MSC-1 monotherapy for further evaluation in the expansion part of the study | Patients will be evaluated for approximately 6 months or until disease progression
  Assessment of frequency & severity of adverse events
Assess the preliminary anti-tumor activity of MSC-1 monotherapy | Patients will be evaluated for approximately 6 months or until disease progression
  Determine objective response rate (ORR)

SECONDARY OUTCOMES:
Confirm safest dose of MSC-1 for further study | Patients will be evaluated for approximately 6 months or until disease progression
  Assessment of adverse events
Characterize the PK of MSC-1 | Patients will be evaluated before and after each dose of MSC-1 for approximately 6 months or until disease progression. PK will be evaluated more frequently for the first 2 cycles of treatment
  Serum levels of MSC-1

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - HonorHealth, Scottsdale, Arizona
  - START MidWest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center- Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center- Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Hospital Universitario Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor Website — http://www.astrazenecaclinicaltrials.com
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=MSC-1-101&attachmentIdentifier=168a4a3e-7b7f-470d-a1b1-fe54d4ba23ff&fileName=MSC-1-101_CSRSynopsis.pdf&versionIdentifier=